CLINICAL TRIAL: NCT00546806
Title: The University Health Network Whiplash Intervention Trial: A Randomized Controlled Trial of the Effectiveness and Cost-effectiveness of Three Programs of Care for the Treatment of Whiplash-associated Disorders
Brief Title: University Health Network Whiplash Intervention Trial
Acronym: WIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AVIVA Canada (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-0623-A
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Whiplash Injuries
Keywords: Rehabilitation,; Treatment outcome,; Whiplash injuries,; Randomized Clinical Trials
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AVIVA "Soft Tissue Injury Care Model"
  Interventions: Other: Programs of Care
- 2 (Experimental): Pre-approved Framework Guideline for Grade I and II Whiplash Associated Disorders (PAF)
  Interventions: Other: Programs of Care
- 3 (Active Comparator): Physician-based Education and Activation
  Interventions: Other: Programs of Care

INTERVENTIONS:
Other: Programs of Care — Two physiotherapy programs of care for the experimental groups; Physician-based education and activation for the active comparator group.

SUMMARY:
Whiplash is the most common traffic injury, affecting 83% of people involved in motor vehicle collisions. People with whiplash injuries often experience pain and disability that can last for a long period. This may subsequently lead to an increased use of the health care system. Preventing chronic symptoms is a priority for clinicians, insurers, and policy makers. However, there are very few factors that can be changed by treatment to prevent prolonged symptoms. Providing effective care at the appropriate time is one aspect that can be changed and needs to be studied. To date, no randomized clinical trials have investigated the effectiveness of multidisciplinary rehabilitation programs for the management of patients with whiplash-associated disorders. Additionally, there is no evidence to suggest whether rehabilitation programs are superior to physician-based care at improving whiplash-associated symptoms. Thus, there is a need for a randomized trial to determine what program results in the best outcomes for patients.

The purpose of this study is to compare three programs of care that are currently available in Ontario for the management of patients with Whiplash-associated disorders.

The results of this study will demonstrate which of three programs of care is superior in improving the physical and mental health of patients with whiplash-associated disorders. The results will help guide the development and implementation of effective and cost-effective programs of care by informing clinicians, insurers and government on the best rehabilitation options for patients with whiplash injuries.

DETAILED DESCRIPTION:
Background: Whiplash is the most common traffic injury, affecting 83% of people involved in motor vehicle collisions. It results in a significant burden of pain, disability and health care utilization. Preventing chronic whiplash is a priority for clinicians, insurers, and policy makers. However, whiplash injuries are resistant to treatment and few of its prognostic factors are modifiable through intervention. One of the rare factors amenable to change is the provision of timely and effective clinical care. To date, no randomized trials that have investigated the effectiveness of a coordinated and staged multidisciplinary rehabilitation program aimed at improving the health outcomes of patients with whiplash-associated disorders. Moreover, it is not known whether rehabilitation programs are superior to physician care in promoting better health outcomes. Overall, there is a need for a pragmatic randomized controlled trial to investigate what program of care yields the best outcomes for patients.

Purpose: To compare the effectiveness and cost-effectiveness of the "Soft Tissue Injury Care Model" designed by AVIVA Canada, the "Pre-approved Framework Guideline for Grade I and II Whiplash Associated Disorders" recommended by the Financial Services Commission of Ontario and a physician-based "Education and Activation" intervention on the rate of self-rated recovery from whiplash-associated disorders.

Methods: We designed a three-arm pragmatic randomized controlled trial. Eligible participants will be randomly allocated to receive one of three program of care: 1) the "Soft Tissue Injury Care Model" designed by AVIVA Canada;2) the "Pre-approved Framework Guideline for Grade I and II Whiplash Associated Disorders" recommended by the Financial Services Commission of Ontario ; or 3) a physician-based "Education and Activation" intervention.

Significance: The results of this study will provide evidence regarding the effectiveness of three commonly used management strategies for whiplash injuries in Ontario. The results will help guide the development of effective and cost-effective programs of care and inform insurance and government policy on the rehabilitation of whiplash injuries.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* make an insurance claim for physical injury within 21 days of the traffic collision
* diagnosed with Grade I or Grade II WAD
* report an average neck pain since the accident of at least 3 on a 0-10 "Numerical Rating Scale"
* able to give written informed consent and complete interviews in English

Exclusion Criteria:

* a fracture/dislocation of the spine or any major bone
* head trauma associated with loss of consciousness
* past whiplash or work-related neck injury within the year prior to their current injury
* active systemic diseases
* previous neck surgery
* received treatment from a physiotherapist or a chiropractor for neck pain in the three months preceding the motor vehicle collision
* individuals who do not reside in the Greater Toronto, Mississauga, Burlington, Cambridge or Kitchener areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2008-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Global perceived recovery, Costs | baseline, 6 weeks, 3, 6, 9 months and 1 year

SECONDARY OUTCOMES:
Neck pain intensity, Whiplash disability, Health-related quality of life, Depressive symptomatology, Satisfaction with care and satisfaction with treatment, Time on insurance benefit, Recurrence, Adverse events | baseline, 6 weeks, 3, 6, 9 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Côté, DC, PhD, Principal Investigator — University Health Network, Toronto
Locations (5):
- Canada (5):
  - Harwood Rehab and Sports Injury Clinic, Ajax, Ontario
  - UHN Rehabilitation Solutions, Cambridge Site, Cambridge, Ontario
  - UHN Rehabilitation Solutions, Mississauga Site, Mississauga, Ontario
  - Pickering Rehab Clinic, Pickering, Ontario
  - UHN Rehabilitation Solutions, Toronto Western Hospital Site, Toronto, Ontario

REFERENCES:
- [Background] Cote P, Cassidy JD, Carette S, Boyle E, Shearer HM, Stupar M, Ammendolia C, van der Velde G, Hayden JA, Yang X, van Tulder M, Frank JW. Protocol of a randomized controlled trial of the effectiveness of physician education and activation versus two rehabilitation programs for the treatment of Whiplash-associated Disorders: The University Health Network Whiplash Intervention Trial. Trials. 2008 Dec 24;9:75. doi: 10.1186/1745-6215-9-75. PMID 19108741
- [Background] van der Velde G, Cote P, Bayoumi AM, Cassidy JD, Boyle E, Shearer HM, Stupar M, Jacobs C, Ammendolia C, Carette S, van Tulder M. Protocol for an economic evaluation alongside the University Health Network Whiplash Intervention Trial: cost-effectiveness of education and activation, a rehabilitation program, and the legislated standard of care for acute whiplash injury in Ontario. BMC Public Health. 2011 Jul 27;11:594. doi: 10.1186/1471-2458-11-594. PMID 21794155
- [Derived] Marchand AA, Hogg-Johnson S, Cote P. Baseline Depressive Symptoms Do Not Moderate the Association Between Baseline Symptom Severity and Time to Recovery in Individuals with Grade I-II Whiplash-Associated Disorders: A Secondary Analysis of a Randomized Controlled Trial. Am J Phys Med Rehabil. 2023 Oct 1;102(10):861-866. doi: 10.1097/PHM.0000000000002223. Epub 2023 Mar 1. PMID 36882302
- [Derived] Cote P, Boyle E, Shearer HM, Stupar M, Jacobs C, Cassidy JD, Carette S, van der Velde G, Wong JJ, Hogg-Johnson S, Ammendolia C, Hayden JA, van Tulder M, Frank JW. Is a government-regulated rehabilitation guideline more effective than general practitioner education or preferred-provider rehabilitation in promoting recovery from acute whiplash-associated disorders? A pragmatic randomised controlled trial. BMJ Open. 2019 Jan 24;9(1):e021283. doi: 10.1136/bmjopen-2017-021283. PMID 30679283